CLINICAL TRIAL: NCT05663866
Title: Subcutaneous Methotrexate, Oral Dexamethasone or Oral Montelukast for the Prevention of Infusion Related Reaction Associated With Amivantamab, an EGFR-MET Bispecific Antibody, Among Post-osimertinib Treated EGFRm NSCLC; SKIPPirr, a Phase 2 Study
Brief Title: Premedication to Reduce Amivantamab Associated Infusion Related Reactions
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109305; 61186372NSC2005 (Other: Janssen Research & Development, LLC); 2022-000974-25 (EudraCT Number); 2023-506578-11-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-12-16; First posted 2022-12-23 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dexamethasone; montelukast; Methotrexate; amivantamab; lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Background Anti-cancer Therapy with Amivantamab Plus Lazertinib (Experimental): Participant will receive following treatments in 4 different cohorts prior to administration of combination therapy of IV Amivantamab and oral Lazertinib (anti-cancer regimen): dexamethasone dose-1 in Cohort A; dexamethasone dose-2 in Cohort A2; montelukast in Cohort B; and methotrexate in Cohort C.
  Interventions: Drug: Dexamethasone; Drug: Montelukast; Drug: Methotrexate; Drug: Amivantamab; Drug: Lazertinib

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be administered orally.
Drug: Montelukast — Montelukast will be administered orally.
Drug: Methotrexate — Methotrexate will be administered subcutaneously.
Drug: Amivantamab — Amivantamab will be administered intravenously.
  Other Names: JNJ-61186372
Drug: Lazertinib — Lazertinib tablets will be administered orally.
  Other Names: JNJ-73841937

SUMMARY:
The purpose of the study is to separately assess the potential of dexamethasone, montelukast and methotrexate administration, prior to amivantamab infusion given through a needle in the vein, to decrease the incidence and/or severity of first-dose infusion related reactions.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have advanced or metastatic non-small cell lung cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* A female participant using oral contraceptives must use an additional barrier contraceptive method
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 3 months after receiving the last dose of study treatment, oral lazertinib and intravenous (IV) Amivantamab
* Each participant, or legally authorized representative, where allowed, must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Progressed on or after prior treatment with osimertinib and platinum-based chemotherapy. Prior use of first-or-second generation epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI) is allowed if administered prior to osimertinib
* Previously identified EGFR-mutated non-small cell lung cancer (NSCLC) (EGFR Exon19 deletion or L858R) (identified locally in a Clinical Laboratory Improvement Amendments [CLIA]-certified laboratory [or equivalent])

Exclusion Criteria:

* Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis
* Prior treatment with anti PD-1 or anti PD-L1 antibody within 6 weeks of planned first dose of study treatment or immune-mediated rash from checkpoint inhibitors that has not resolved prior to enrollment
* Participant has symptomatic brain metastases. A participant with asymptomatic or previously treated and stable brain metastases may participate in this study. Participants who have completed definitive therapy, are not on steroids, and have a stable clinical status for at least 2 weeks prior to study treatment are allowed. If brain metastases are diagnosed on Screening imaging, the participant may be enrolled, or rescreened for eligibility, after definitive treatment if above criteria are met
* Any toxicities from prior anticancer therapy must have resolved to common terminology criteria for adverse events (CTCAE) version 5.0 Grade 1 or baseline level (except for alopecia [any grade], Grade less than or equal to [<=] 2 peripheral neuropathy, and Grade <=2 hypothyroidism stable on hormone replacement therapy)
* Prior treatment with amivantamab or lazertinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2026-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (36):
- United States (3):
  - Compassionate Cancer Care, Fountain Valley, California
  - Virginia Cancer Specialists, Fairfax, Virginia
  - UW Medicine Valley Medical Center, Renton, Washington
- France (6):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - Centre Leon Berard, Lyon
  - Hopital Cochin, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - CHU Rouen Hopital Charles Nicolle, Rouen
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
- Spain (14):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp. San Pedro de Alcantara, Cáceres
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Inst. Valenciano de Oncologia, Valencia
  - Hosp. Gral. Univ. Valencia, Valencia
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Medical Center, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Dexamethasone 4 Milligrams (mg): Participants were administered with oral dexamethasone 4 mg tablet as a prophylactic treatment twice a day (8 mg total daily dose) on Day -1 (Cycle 1) prior to combination therapy of lazertinib 240 mg oral tablets and IV infusion of amivantamab 1050 mg (for participants less than [<] 80 kilograms [kg]) or 1400 mg (for participants greater than or equal to [>=] 80 kg) on Cycle 1 Day 1 until disease progression or withdrawal from study. Each cycle was of 28 days.
- Cohort A2: Dexamethasone 8 mg: Participants were administered with oral dexamethasone 8 mg tablet as a prophylactic treatment twice a day (16 mg total daily dose) on Day -2 and -1 (Cycle 1) and 8 mg approximately one hour prior to IV infusion of amivantamab 1050 mg (for participants <80 kg) or 1400 mg (for participants >=80 kg) on Cycle 1 Day 1 until disease progression or withdrawal from study. Each cycle was of 28 days.
- Cohort B: Montelukast 10 mg: Participants were administered with oral montelukast 10 mg tablet as a prophylactic treatment once daily in the morning on Days - 4, -3, -2, -1, and Cycle 1 Day 1 prior to combination therapy of lazertinib 240 mg oral tablets and IV infusion of amivantamab 1050 mg (for participants <80 kg) or 1400 mg (for participants >=80 kg) on Cycle 1 Day 1 until disease progression or withdrawal from study. Each cycle was of 28 days.
- Cohort C: Methotrexate 25 mg: Participants were administered with a single dose of methotrexate 25 mg subcutaneous injection as a prophylactic treatment on any day between Days -7 and Day -3 (Cycle 1) prior to combination therapy of lazertinib 240 mg oral tablets and IV infusion of amivantamab 1050 mg (for participants <80 kg) or 1400 mg (for participants >=80 kg) on Cycle 1 Day 1 until disease progression or withdrawal from study. Each cycle was of 28 days.
Period: Overall Study
Arm/Group | Cohort A: Dexamethasone 4 Milligrams (mg) | Cohort A2: Dexamethasone 8 mg | Cohort B: Montelukast 10 mg | Cohort C: Methotrexate 25 mg
Started | 6 | 41 | 15 | 6
Completed | 0 | 4 | 2 | 0
Not Completed | 6 | 37 | 13 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 2
Not completed — Progressive disease | 4 | 8 | 5 | 2
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Ongoing | 1 | 27 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Dexamethasone 4 Milligrams (mg) | Cohort A2: Dexamethasone 8 mg | Cohort B: Montelukast 10 mg | Cohort C: Methotrexate 25 mg | Total
Number analyzed (Participants) | 6 | 41 | 15 | 6 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (13.60) | 62.0 (9.68) | 65.0 (8.72) | 66.2 (11.96) | 62.7 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 26 | 10 | 5 | 44
  Male | 3 | 15 | 5 | 1 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 0 | 6
  Not Hispanic or Latino | 3 | 31 | 13 | 6 | 53
  Unknown or Not Reported | 1 | 8 | 0 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 24 | 10 | 6 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 4 | 10 | 4 | 0 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Infusion-related Reactions (IRRs) at Cycle 1 Day 1
Description: Percentage of participants with IRRs at Cycle 1 Day 1 was reported. IRRs were defined as IRR events with onset time within 24 hours of the start of the first amivantamab infusion and prior to the start of amivantamab infusion on Cycle 1 Day 2. IRR included chills, dyspnea, flushing, nausea, chest discomfort, vomiting, tachycardia, hypotension, and fever. IRRs that occurred on Cycle 1 Day 2 pre-infusion were considered under Cycle 1 Day 1.
Time Frame: Cycle 1 Day 1 (each cycle of 28 days)
Population: The per protocol analysis set included all participants who had received all prophylaxis treatment based on schedule and had received the administration of amivantamab and lazertinib on Cycle 1 Day 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Dexamethasone 4 Milligrams (mg) | Cohort A2: Dexamethasone 8 mg | Cohort B: Montelukast 10 mg | Cohort C: Methotrexate 25 mg
Number analyzed (Participants) | 6 | 40 | 15 | 6
Percentage of participants | 83.3 [35.9 to 99.6] | 22.5 [10.8 to 38.5] | 66.7 [38.4 to 88.2] | 83.3 [35.9 to 99.6]

2. Secondary Outcome: Percentage of Participants With Adverse Events of Infusion-related Reactions (IRRs) During Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2027-07

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) of Infusion-related Reactions (IRRs) as Per Severity up to End of Cycle 3 (Cycle 3 Day 28)
Time Frame: From Cycle 1 Day 1 up to Cycle 3 Day 28 (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2027-07

4. Secondary Outcome: Percentage of Participants With IRRs up to End of Treatment (EOT)
Time Frame: From Cycle 1 Day 1 (each cycle of 28 days) up to 27.3 months
Reporting Status: Not Posted, anticipated posting 2027-07

5. Secondary Outcome: Percentage of Participants With Other Adverse Events (AEs): Non-IRRs
Time Frame: From Cycle 1 Day 1 (each cycle of 28 days) up to 28.3 months
Reporting Status: Not Posted, anticipated posting 2027-07

6. Secondary Outcome: Duration of Infusion Time for Pre-amivantamab Infusion Medications, IV Amivantamab Infusion, and Post-amivantamab Infusion Medications on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2027-07

7. Secondary Outcome: Percentage of Participants Completing Amivantamab Infusion Within 4 Hours on Cycle 1 Day 1
Time Frame: Up to 4 hours on Cycle 1 Day 1 (each cycle of 28 days)
Reporting Status: Not Posted, anticipated posting 2027-07

8. Secondary Outcome: Overall Response Rate (ORR)
Time Frame: From Cycle 1 Day 1 (each cycle of 28 days) up to 28.3 months
Reporting Status: Not Posted, anticipated posting 2027-07

9. Secondary Outcome: Duration of Response (DOR)
Time Frame: From Cycle 1 Day 1 (each cycle of 28 days) up to 28.3 months
Reporting Status: Not Posted, anticipated posting 2027-07

ADVERSE EVENTS:
Time Frame: From Cycle 1 Day 1 up to 10 months (each cycle of 28 days)
Description: Safety analysis set included all participants who received at least 1 administration of amivantamab and lazertinib. The study was to evaluate reduction in infusion-related reactions (IRRs) associated with amivantamab when given after prophylactic treatment with dexamethasone, montelukast, and methotrexate. Hence, safety data was collected and analyzed only for amivantamab/ amivantamab + lazertinib and is reported below.
Groups:
- Cohort A1: Dexamethasone 4 Milligrams (mg): Participants were administered with oral dexamethasone 4 mg tablet as a prophylactic treatment twice a day (8 mg total daily dose) on Day -1 (Cycle 1) prior to combination therapy of lazertinib 240 mg oral tablets and IV infusion of amivantamab 1050 mg (for participants less than [<] 80 kilograms [kg]) or 1400 mg (for participants greater than or equal to [>=] 80 kg) on Cycle 1 Day 1 until disease progression or withdrawal from study. Each cycle was of 28 days.
Arm/Group | Cohort A1: Dexamethasone 4 Milligrams (mg) | Cohort A2: Dexamethasone 8 mg | Cohort B: Montelukast 10 mg | Cohort C: Methotrexate 25 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 4/41 | 2/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 20/41 | 5/15 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 41/41 | 15/15 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Dexamethasone 4 Milligrams (mg) (N=6) | Cohort A2: Dexamethasone 8 mg (N=41) | Cohort B: Montelukast 10 mg (N=15) | Cohort C: Methotrexate 25 mg (N=6)
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia Aspiration (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 2 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Abnormal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Dexamethasone 4 Milligrams (mg) (N=6) | Cohort A2: Dexamethasone 8 mg (N=41) | Cohort B: Montelukast 10 mg (N=15) | Cohort C: Methotrexate 25 mg (N=6)
Rash (Skin and subcutaneous tissue disorders) | 2 | 17 | 8 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5 | 3 | 4
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 | 7 | 3 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 6 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 10 | 6 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 14 | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 8 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 2 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 4 | 2 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 2 | 16 | 10 | 2
Covid-19 (Infections and infestations) | 0 | 1 | 5 | 0
Folliculitis (Infections and infestations) | 0 | 3 | 3 | 0
Conjunctivitis (Infections and infestations) | 0 | 3 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Eye Infection (Infections and infestations) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Rash Pustular (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 9 | 5 | 0
Asthenia (General disorders) | 2 | 7 | 3 | 0
Chills (General disorders) | 2 | 0 | 6 | 2
Chest Discomfort (General disorders) | 0 | 1 | 2 | 4
Fatigue (General disorders) | 0 | 3 | 3 | 1
Pyrexia (General disorders) | 1 | 1 | 2 | 1
Malaise (General disorders) | 0 | 2 | 1 | 0
Infusion Site Extravasation (General disorders) | 0 | 1 | 1 | 0
Feeling Hot (General disorders) | 1 | 0 | 0 | 0
Lithiasis (General disorders) | 0 | 0 | 0 | 1
Localised Oedema (General disorders) | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
Temperature Regulation Disorder (General disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 5 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 17 | 4 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 4 | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 8 | 4 | 1
Headache (Nervous system disorders) | 0 | 8 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 3
Paraesthesia (Nervous system disorders) | 1 | 3 | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 2 | 1 | 1
Petit Mal Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 8 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 2 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 5 | 2 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 5 | 2 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 2 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 2 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 1 | 0
Blood Creatine Increased (Investigations) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 1 | 0
Dry Eye (Eye disorders) | 0 | 2 | 1 | 0
Trichiasis (Eye disorders) | 0 | 0 | 1 | 1
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 2 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Ear Inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Genital Rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT05663866/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT05663866/SAP_001.pdf